CLINICAL TRIAL: NCT02741882
Title: Rash Accompanied by Three or More Dengue-like Symptoms During Pregnancy and Microcephaly: Case-control Study
Brief Title: Zika and Microcephaly: Case-control Study
Status: Completed | Type: Observational
Sponsor: Laboratório Sabin (Industry)
Responsible Party: Principal Investigator, Gustavo Barcelos Barra, Pharm.D Ph.D, Laboratório Sabin
Other Study IDs: Zika and microcephaly
Record Dates: First submitted 2016-04-13; First posted 2016-04-18 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Microcephaly
Keywords: Microcephaly; zika Virus; Case-control study
MeSH Terms: conditions — Microcephaly; Zika Virus Infection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cases: Mothers who delivered a baby with microcephaly at Nossa Senhora de Lourdes maternity hospital located in Aracaju, state of Sergipe, Brazil from September 1, 2015 through January 5, 2016. The intervention will be a questionary.
  Interventions: Other: Questionary
- Controls: Mothers who delivered a baby without microcephaly at Nossa Senhora de Lourdes maternity hospital located in Aracaju, state of Sergipe, Brazil from September 1, 2015 through January 5, 2016. The intervention will be a questionary.
  Interventions: Other: Questionary

INTERVENTIONS:
Other: Questionary — Questionary with clinical, demographic and behavior outcomes at the pregnancy period

SUMMARY:
It is suspected that zika virus infection during pregnancy is associated with microcephaly. The objective of this study is to investigate the occurrence of rash accompanied by three or more dengue-like signs and symptoms during pregnancy is related to the microcephaly using the case-control design.

DETAILED DESCRIPTION:
The investigators will carry out a case-control study among mothers who delivered their babies at Nossa Senhora de Lourdes maternity hospital located in Aracaju, state of Sergipe, Brazil from September 1, 2015 through January 5, 2016. Data sources for the phase I of the study will consist of medical records review and a standard questionnaire applied by telephone to collect information about demographic features, clinical signs and symptoms, and the duration and severity of the illness. Phase II will include dengue, chikungunya and dengue serologic test results as secondary outcome, if available. The objective of this study is to investigate the occurrence of rash accompanied by three or more dengue-like signs and symptoms during pregnancy is related to the microcephaly using the case-control design

ELIGIBILITY:
Inclusion Criteria:

* Delivered a baby at nossa senhora de lourdes maternity from September 1, 2015 through january 5, 2016.

Exclusion Criteria:

* Syphilis during pregnancy, toxoplasmosis during pregnancy, consanguinity, other genetics disorder, alcohol or abuse drug consumption during pregnancy.

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Mothers who delivered their babies at Nossa Senhora de Lourdes maternity hospital located in Aracaju, state of Sergipe, Brazil from September 1, 2015 through January 5, 2016.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2016-02; Primary Completion 2016-08 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Zika virus infection clinical outcomes during pregnancy | From September 1, 2015 through January 5, 2016
  acute onset of generalized rash together with three of the following symptoms: Conjunctivitis, arthralgia, mild-fever or periarticular edema.

SECONDARY OUTCOMES:
zika virus serology | march, 2016 through July 5, 2016
  If available, zika virus serology will be performed
Chikungunya virus serology | march, 2016 through July 5, 2016
  If available, chikungunya virus serology will be performed
Dengue virus serology | march, 2016 through July 5, 2016
  If available, Dengue virus serology will be performed

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo B Barra, ph.D, Principal Investigator — Sabin Laboratory
Locations (1):
- Sabin laboratory, Brasília, Federal District, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Santa Rita TH, Barra RB, Peixoto GP, Mesquita PG, Barra GB. Association between suspected Zika virus disease during pregnancy and giving birth to a newborn with congenital microcephaly: a matched case-control study. BMC Res Notes. 2017 Sep 6;10(1):457. doi: 10.1186/s13104-017-2796-1. PMID 28877754